CLINICAL TRIAL: NCT03708562
Title: everlinQ Endovascular Access Systems Enhancements (EASE-2) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-0038
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Results first posted 2020-01-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoAVF (Other)
  Interventions: Device: everlinQ endoAVF System

INTERVENTIONS:
Device: everlinQ endoAVF System — The everlinQ device is a single-use disposable device. The everlinQ catheter system consists of two flexible, magnetic catheters. Once the catheters are properly inserted and aligned, the magnets contained in each catheter attract to one another, approximating the vessels while simultaneously aligning the electrode with the backstop. Radiofrequency (RF) energy is delivered to the electrode whereby the arterio-venous fistula (AVF) is created.

SUMMARY:
Prospective, single-center study to evaluate the everlinQ endoAVF System when used to create an endoAVF in hemodialysis patients. This study aims to investigate expansion of the percutaneous venous access location to the superficial system which may provide additional procedural benefit.

DETAILED DESCRIPTION:
A total of up to 50 subjects will be enrolled and will undergo an endoAVF creation procedure using the everlinQ System. All subjects may be followed for up to 12 months post index procedure based on Investigator's discretion. The duration of the study is expected to be approximately two (2) years.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for a native arteriovenous fistula.
2. Adult (age >18 years old).
3. Established, non-reversible kidney failure requiring hemodialysis (including pre-dialysis patients).
4. Target vein diameter(s) at fistula site ≥ 2.0 mm.
5. Target artery diameter at fistula site ≥ 2.0 mm.
6. Procedural access site artery and vein diameter ≥ 2.0 mm.
7. At least one superficial outflow vein diameter ≥ 2.5 mm and in communication with the perforating vein.
8. Estimated life expectancy > 1 year.
9. Patient is free of clinically significant conditions or illness within 30 days prior to the AV fistula that may compromise the procedure.
10. Presence of an antecubital perforating vein diameter ≥ 2.0 mm.

Exclusion Criteria:

1. Known central venous stenosis or central vein narrowing > 50% based on imaging on the same side as the planned AVF creation.
2. Upper extremity venous occlusion(s) and/or vessel abnormality(ies) on the same side as the planned AVF creation that precludes endovascular AVF creation by the everlinQ System as deemed by the interventionalists' clinical judgment.
3. Prior surgically created access in the planned treatment location.
4. Functioning surgical access in the planned treatment arm.
5. Pregnant women.
6. New York Heart Association (NYHA) class III or IV heart failure.
7. Hypercoagulable state.
8. Known bleeding diathesis.
9. Immunosuppression, defined as use of immunosuppressive medications used to treat an active condition.
10. Documented history of drug abuse including intravenous drugs within six months of AVF creation.
11. "Planned" concomitant major surgical procedure within 6 months of enrollment or previous major surgery within 30 days of enrollment.
12. Currently being treated with another investigational device or drug.
13. Known allergy to contrast dye which cannot be adequately pre-medicated.
14. Known adverse effects to sedation and/or anesthesia which cannot be adequately pre- medicated.
15. Patients who do not have an ulnar or radial artery.
16. Distance between target artery and vein or other anatomical abnormality will not permit catheters to be introduced, navigated to fistula site, or allow magnets to align vessels sufficiently to create the fistula.
17. Evidence of calcification in vessels at the fistula site.
18. Evidence of active infections on the day of the index procedure.
19. Written informed consent not obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, Principal Investigator — Sanatorio Italiano, Paraguay
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The EverlinQ Endovascular Access Systems Enhancements (EASE-2) study began enrollment on October 5th 2017 and the last patient was enrolled on May 23rd 2018.
Period: Overall Study
Arm/Group | endoAVF
Started | 24
Completed | 12
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- endoAVF: everlinQ endoAVF System: The everlinQ device is a single-use disposable device. The everlinQ catheter system consists of two flexible, magnetic catheters. Once the catheters are properly inserted and aligned, the magnets contained in each catheter attract to one another, approximating the vessels while simultaneously aligning the electrode with the backstop. RF energy is delivered to the electrode whereby the arterio-venous fistula (AVF) is created.
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Paraguay | 24
Access Artery [Count of Participants; unit: Participants]
  Brachial | 2
  Ulnar | 16
  Radial | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedural Success
Description: Procedure Success was defined as successful endoAVF creation confirmed via intraprocedural angiography/fistulogram or duplex ultrasound verification performed post procedure.
Time Frame: At time of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Participants | 19

2. Primary Outcome: Adverse Event Rate
Description: Percentage of patients who experience one or more adverse events during the first 3 months following successful endoAVF creation. Adverse events were site-reported and reviewed by an independent Medical Monitor and the Clinical Events Committee (CEC).
Time Frame: 3 months following endoAVF creation
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Participants | 4

3. Secondary Outcome: Percentage of Participants With Primary Patency at 6 Months Post Index Procedure
Description: Primary Patency was defined as the time interval between the endoAVF index procedure and the earlier of a) any intervention designed to maintain or reestablish patency, b) access thrombosis, or c) access abandonment. Kaplan-Meier (KM) was used to analyze the data.
Time Frame: 6 months post index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Percentage of participants | 70.8

4. Secondary Outcome: Number of Participants With EndoAVF Maturation at 1, 3, and 6 Months Post Index Procedure
Description: Maturity of the endoAVF was defined by duplex ultrasound criteria, as described in the literature as a useful surrogate of suitability for dialysis. Maturation was defined as duplex ultrasound flow in the brachial artery of at least 500 ml/min and a vein diameter ≥ 4mm, without significant stenosis or thrombosis. If a subject was on hemodialysis, maturity was defined by successful dialysis with 2-needles at least once.
Time Frame: 1, 3, and 6 months post index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Participants
  1 month post index procedure | 19
  3 months post index procedure | 20
  6 months post index procedure | 20

5. Secondary Outcome: Time to Cannulation (Months)
Description: The interval of time from the index procedure to successful 2-needle cannulation of the endoAVF.
Time Frame: Months from index procedure to cannulation
Population: Analysis population is lower than total subject number due to subject withdrawals before this endpoint could be analyzed.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | endoAVF
Number analyzed (Participants) | 13
Months | 1.2 (0.3)

6. Secondary Outcome: Number of Participants With Cannulation Success at Defined Follow-up Intervals
Description: A subject was referred to as a 'cannulation success' with the first successful 2-needle cannulation of the endoAVF access circuit. "Cannulation Success" was defined by at least one successful hemodialysis session through a 2-needle cannulation of the endoAVF access circuit. "Cumulative Cannulation Success" = (Successes Through End Current Interval) / (Subjects on Dialysis at Start Current Interval + Censored Dialysis Subjects through End of Last Interval).
Time Frame: 0-10 days, 11-45 days, 46-135 days, 136-210 days post index procedure
Population: Overall number of participants analyzed (n), and participants analyzed for each follow-up period varies from total participants in the study (N=24) according to the number of participants that attend follow-up and/or had data relevant to the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 20
Participants
  0 to 10 days post index procedure: number analyzed (Participants) | 17
  0 to 10 days post index procedure | 0
  11 to 45 days post index procedure: number analyzed (Participants) | 19
  11 to 45 days post index procedure | 11
  46-135 days post index procedure | 13
  136-210 days post index procedure | 13

7. Secondary Outcome: Percentage of Participants With Assisted Primary Patency at 6 Months
Description: Defined as the interval from access placement to thrombosis or abandonment; not triggered by access circuit interventions performed in the absence of occlusion.
Time Frame: 6 months post index procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Percentage of Participants | 70.8

8. Secondary Outcome: Percentage of Participants With Secondary Patency at 6 Months Post Index Procedure
Description: Secondary Patency was defined as the time interval between the endoAVF index procedure and a) access abandonment, or b) loss to thrombosis, irrespective of intervening surgical or endovascular interventions designed to re-establish functionality in a stenosed or thrombosed access circuit.
Time Frame: 6 months post index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Percentage of participants | 70.8

9. Secondary Outcome: Percentage of Participants With Functional Patency of the endoAVF at 6 Months Post Index Procedure
Description: The interval of time from the first 2-needle dialysis utilizing the access until access abandonment (SVS Reporting Standards definition). Functional Patency was the interval of time from the first 2-needle dialysis of the endoAVF access circuit until access abandonment.
Time Frame: 6 months post index procedure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Percentage of participants | 90.9 [50.8 to 98.7]

10. Secondary Outcome: Number of Participants With EndoAVF Related Reintervention
Description: The re-intervention rate for endoAVF (defined as any intervention required to maintain or re-establish patency) was calculated at each available follow-up visit post index procedure.
Time Frame: At 6 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Participants | 3

11. Secondary Outcome: Percentage of Participants With Modified Primary Patency at 6 Months Post Index Procedure
Description: Modified Primary Patency was defined as a measure of patency that, in addition to occlusion or reinterventions within the access circuit, also included coil embolization or open surgical ligation of outflow venous branches as failures of patency when they occur after the index procedure.
Time Frame: 6 months post index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 24
Percentage of participants | 70.8

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were collected through 6-months post-index procedure.
Description: Significant Events were classified by the independent Medical Monitor and included device or procedure-related adverse events that either a) could be limb-threatening if not promptly identified or treated, or b) required additional therapy to reestablish patency of the endoAVF access circuit, irrespective of whether they met the criteria for an SAE.
Arm/Group | endoAVF
All-Cause Mortality (participants affected / at risk) | 2/24
Serious Adverse Events (participants affected / at risk) | 4/24
Other Adverse Events (participants affected / at risk) | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | endoAVF (N=24)
Thrombosis (Vascular disorders) | 2 (2)
Pseudoanurysm (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | endoAVF (N=24)
Pseudo-aneurysm (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)
Occlusion (Vascular disorders) | 1 (1)
Swelling (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT03708562/Prot_SAP_000.pdf